CLINICAL TRIAL: NCT01946828
Title: Evaluation of the FIM - a Non Invasive Device for Temporarily and Quick Pupil Dilation (Mydriasis)
Acronym: TP 7601-CL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TASMC-13-AM-0280-CTIL
Record Dates: First submitted 2013-09-11; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Pupil Dilation
Keywords: Field Induced Mydriasis; FIM; ATI
MeSH Terms: conditions — Mydriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FIM (Experimental): safety and efficacy of the FIM when exposed to a large and varied population of patients and users and operated according to its instructions for use
  Interventions: Device: FIM

INTERVENTIONS:
Device: FIM — Field Induced Mydriasis device

SUMMARY:
The objective of this clinical trial is to evaluate the FIM optimal configuration and confirm the safety and performance/efficacy of the FIM when exposed to a larger and more varied population of users.

DETAILED DESCRIPTION:
70 Eligible subjects will be enrolled to the study and examined with the FIM to determine the degree of pupil dilation/Contraction resistance.

The study will be conducted in two main stages: 1) pupil dilation measuring and 2) functional examination. The tests' sequence will be randomized, at least 30 minutes between each test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and not diagnosed with any chronic disease that might influence the eye and pupilary muscle.
* Age 18-45 years old.
* Willing and able to sign the informed consent, after reading the study information form

Exclusion Criteria:

* Any known or diagnosed neurological disorders.
* A known medical history of ophthalmic surgery or any other disease that might influence the iris control muscle.
* Volunteers with a narrow or closed angle of the anterior chamber
* Presence of a corneal pathology which precludes measurement of the pupil dilatation
* Using of psychiatric medications
* Pregnancy
* Recent use (last 48hr) of pupil dilator eye drops.
* The volunteer is participating in other trials using drugs or devices
* Drug or alcohol abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Safety | 4 months
  number, severity and causality of unexpected, device related adverse events
Functionality | 4 months
  Functionality - ability to perform standard ophthalmologic examination

SECONDARY OUTCOMES:
Usability | 4 months
  Device usability and user satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- See also: ATI Advanced Medical Technologies — http://www.ati-amt.com